CLINICAL TRIAL: NCT04048278
Title: Lidocaine Infusion in Pancreatic Cancer: Translational Studies in a Preclinical Model And Human Subjects
Brief Title: Lidocaine Infusion in Pancreatic Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Effrossyni Votta-Velis, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-1365
Record Dates: First submitted 2019-06-18; First posted 2019-08-07 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-11

CONDITIONS: Pancreatic Cancer
Keywords: Pancreas; Pancreatic Cancer; Lidocaine; Enzymatic Activity; Cytokines; Chemokines; Gene Expression
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Lidocaine; Saline Solution; Injections; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: A prospective randomized placebo-controlled double blinded trial design will be used for the proposed study.
Who Masked: Participant, Care Provider
Masking Description: Both patients and the physicians performing the cases will be unaware of who receives lidocaine or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lidocaine Hydrochloride (Experimental): The IV bolus and infusions of lidocaine to those patients assigned to the lidocaine group will be started in the operating room and will continue until 24 h later. The group receiving the lidocaine infusion will first be administered a 1.0 - 1.5 mg/kg loading infusion over 5 minutes followed by a 1.0 - 1.5 mg/kg/h infusion for 24 h
  Interventions: Drug: Lidocaine Hydrochloride
- Saline Solution for Injection (Placebo Comparator): The group receiving the saline infusion will be administered an equivalent volume of saline infused over 5 min followed by a saline infusion at the same flow rate as that used in the lidocaine group for 24 h (1.0 - 1.5 mg/kg/hr)
  Interventions: Drug: Saline Solution for Injection

INTERVENTIONS:
Drug: Lidocaine Hydrochloride — IV Lidocaine a 1.0 - 1.5 mg/kg loading infusion for perioperative pain control
  Other Names: Xylocaine
  Arms: Lidocaine Hydrochloride
Drug: Saline Solution for Injection — IV Saline a 1.0 - 1.5 mg/kg loading infusion for perioperative pain control
  Other Names: Sodium Chloride
  Arms: Saline Solution for Injection

SUMMARY:
This study elucidates the effects of the intravenous (IV) lidocaine infusion on the biology of pancreatic circulating tumor cells (CTCs) isolated from patients undergoing robotic pancreatectomy for all types of pancreatic cancer.

A prospective randomized controlled double blinded trial design will be used for the proposed study.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the effect of IV lidocaine infusion on various enzymatic activities and associated pathways in isolated CTCs as well as the number of CTCs during the perioperative period in patients undergoing robotic pancreatectomy for pancreatic cancer. It is expected that by downregulating the pathways by lidocaine might affect the enzymatic activity in those CTCs as well as the number of CTCs in the circulation.

A prospective randomized controlled double blinded trial design will be used for the proposed study.

Patients undergoing robotic pancreatectomy for pancreatic cancer will be randomized (ratio 1:1) into two groups: one group will receive a 24-h normal saline infusion and the second group will receive a 24-h lidocaine infusion. Blood samples will be collected in different times perioperatively in order to evaluate the objectives of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Has histologically or cytologically confirmed adenocarcinoma of the pancreas that is considered resectable as well as other types of pancreatic cancer (malignant endocrine and exocrine tumors)
2. Has measurable disease, defined as at least 1 tumor that fulfills the criteria
3. Patients diagnosed with resectable cancer, but upon initial phase of surgical exploration found to have metastatic disease
4. Has read, understood and signed the informed consent form (ICF) approved by the Independent Review Board/Independent Ethics Committee (IRB/IEC)
5. Prior systemic treatments for metastatic disease are permitted, including targeted therapies, biologic response modifiers, chemotherapy, hormonal therapy, or investigational therapy.

Exclusion Criteria:

1. Has American Society of Anesthesiologists (ASA) physical status > 3
2. Has hypersensitivity or allergy to amide-linked local anesthetics
3. Has a second or third degree heart block
4. Has severe sinoatrial block
5. Is currently being treated with any of the following class I antiarrhythmic drugs; quinidine, flecainide, disopyramide, or procainamide
6. Has been treated with amiodarone in the past
7. Has Adams-Stoke syndrome
8. Has Wolff-Parkinson-White syndrome
9. Has a history of blood clots, pulmonary embolism, or deep vein thrombosis unless controlled by anticoagulant treatment
10. Has a known history of human immunodeficiency virus (HIV) positivity or untreated and uncontrolled hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2018-11-08 (Actual); Primary Completion 2025-11-08 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Specimen outcome measure. | Outcomes will be evaluated perioperatively
  Src Tyrosine Kinase Enzymatic activity in CTCs. Fluorescence intensity will be used to measure Src phosphorylation in circulating tumor cells.
Specimen outcome measure. | Outcomes will be evaluated perioperatively
  Cytokine Levels in Serum (pg/ml)
Specimen outcome measure. | Outcomes will be evaluated perioperatively
  Chemokine levels in serum (pg/ml)
Upregulation or Downregulation of Gene Expression. | Outcomes will be evaluated perioperatively
  Upregulation or downregulation of gene expression will be measured with the Real Time (RT) square Profiler Polimerase Chain Reaction (PCR )Array Analysis, and Real Time PCR

SECONDARY OUTCOMES:
Specimen outcome measure | Perioperatively
  CTCs Enumeration

CONTACTS AND LOCATIONS:
Overall Officials: Gina E. Votta-Velis, MD PhD, Principal Investigator — Associate Professor
Locations (1):
- University of Illnois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shakhar G, Ben-Eliyahu S. Potential prophylactic measures against postoperative immunosuppression: could they reduce recurrence rates in oncological patients? Ann Surg Oncol. 2003 Oct;10(8):972-92. doi: 10.1245/aso.2003.02.007. PMID 14527919
- [Background] Mokbel K, Choy C, Engledow A. The effect of surgical wounding on tumour development. Eur J Surg Oncol. 2000 Mar;26(2):195. doi: 10.1053/ejso.1999.0771. No abstract available. PMID 10744945
- [Background] Missair A, Cata JP, Votta-Velis G, Johnson M, Borgeat A, Tiouririne M, Gottumukkala V, Buggy D, Vallejo R, Marrero EB, Sessler D, Huntoon MA, Andres J, Casasola OL. Impact of perioperative pain management on cancer recurrence: an ASRA/ESRA special article. Reg Anesth Pain Med. 2019 Jan;44(1):13-28. doi: 10.1136/rapm-2018-000001. PMID 30640648
- [Background] Han L, Chen W, Zhao Q. Prognostic value of circulating tumor cells in patients with pancreatic cancer: a meta-analysis. Tumour Biol. 2014 Mar;35(3):2473-80. doi: 10.1007/s13277-013-1327-5. Epub 2013 Nov 12. PMID 24218336